CLINICAL TRIAL: NCT03779152
Title: Regulation of CCL18 by Corticosteroids in Severe Asthma
Acronym: CCL18
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/0813; 2008-A00370-55 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- non asthmatic subjects
- intermittent asthmatics
- severe asthmatics sensitive to corticosteroids
- severe asthmatics resistant to corticosteroids
- moderate asthmatics

SUMMARY:
The majority of asthmatic patients are well controlled by inhaled corticosteroid treatment, however some severe asthma resist this treatment. CCL18 is a target gene for corticosteroids and its dysfunction may correlate with phenotypes of asthma.

ELIGIBILITY:
Inclusion Criteria:

1. control subjects =

   * non-atopic and non-smoking
   * cutting to negative pneumoallergens,
   * Total IgE levels less than 100 ku / L
   * no clinical history of asthma
   * without background treatment
2. patients with intermittent asthma =

   * being asymptomatic between asthma attacks,
   * with symptoms less than once a week
   * having a forced expiratory volume per second (FEV1) of at least 80% of the theoretical.
   * treated by ß2 mimetics on demand and will not have inhaled corticosteroids.
3. severe asthma insensitive to corticosteroid therapy =

   * continuous or nearly continuous treatment with oral corticosteroids (≥ 50% of the year) / or treatment with IC ≥ 1500 microg beclomethasone dipropionate equivalent (BDP)] airway obstruction fixed with FEV1 ranging from less than 15% after 7 days of oral corticosteroid therapy to 40 mg / day of prednisolone;
   * Followed at the immunoallergology pneumology consultation for at least 1 year will be recruited.
4. Severe corticosensitive asthma = continuous or near continuous treatment with oral corticosteroids (≥ 50% of the year) / or treatment with IC ≥ 1500 microg beclomethasone dipropionate equivalent (BDP)]

   * reversibility of FEV1 after treatment with oral corticosteroids.
   * Followed at the immunoallergology pneumology consultation for at least 1 year will be recruited.
5. controlled moderate asthma treated with inhaled corticosteroids <1500μg equivalent of beclomethasone dipropionate and with: ß2 long-acting mimetics (or anti-leukotriene, or theophylline) for at least 6 months.

Exclusion Criteria:

* existence of a chronic inflammatory pathology other than asthma
* active smoking
* pregnant or lactating women
* have received oral corticosteroid treatment in the previous 3 weeks,
* have received non-steroidal anti-inflammatory drugs (NSAIDs) in the previous 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients consulting for either asthma or chronic rhinitis and meeting the criteria of the control group.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Correlation between CCL18 rate and asthma phenotypes by elisa test | Baseline: one session

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Wallaert, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Calmette, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No